CLINICAL TRIAL: NCT05245656
Title: A Randomized Phase II Trial Comparing Rituximab/Bendamustine(RB) Alternating With Rituximab/Bendamustine/Cytarabine(RBAC) With RB as Induction Therapy in Elderly Patients With Newly Diagnosed and Transplant-ineligible Mantle Cell Lymphoma
Brief Title: A Study Comparing Rituximab/Bendamustin(RB) Alternating With Rituximab/Bendamustin/Cytarabin(RBAC) With RB Therapy in Elderly Patients With Mentle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kim, Seok Jin (Other)
Responsible Party: Sponsor-Investigator, Kim, Seok Jin, Principal Investigator, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-11-126
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RB/RBAC alternating (Experimental): Every 4 weeks for 6 cycles
  RB (1st, 3rd, and 5th cycles)
  * Rituximab + Bendamustine
  RBAC (2nd, 4th, and 6th cycles)
  * Rituximab + Bendamustine + Cytarabine
  Interventions: Drug: RB/RBAC alternating
- RB (Active Comparator): Every 4 weeks for 6 cycles
  - Rituximab + Bendamustine
  Interventions: Drug: RB

INTERVENTIONS:
Drug: RB/RBAC alternating — Patients assigned to the RB alternating with RBAC arm will receive six cycles of alternating RB (odd cycles) or RBAC (even cycles)
  RB (1st, 3rd, and 5th cycles)
  * Rituximab 375mg/m2, IV, D1
  * Bendamustine 90mg/m2, IV, D1-2
  RBAC (2nd, 4th, and 6th cycles)
  * Rituximab 375mg/m2, IV, D1
  * Bendamustine 70mg/m2, IV, D2-3
  * Cytarabine 500mg/m2, IV, D2-4
  Arms: RB/RBAC alternating
Drug: RB — Every 4 weeks for 6 cycles
  * Rituximab 375mg/m2, IV, D1
  * Bendamustine 90mg/m2, IV, D1-2
  Arms: RB

SUMMARY:
This is a phase 2, multicenter, open-label, active-controlled randomized trial to determine efficacy and safety of rituximab/bendamustine (RB) alternating with rituximab/bendamustine/cytarabine (RBAC) compared with standard RB alone in the first-line treatment of elderly patients with mantle cell lymphoma, who are not eligible for high-dose therapy followed by autologous stem cell transplantation.

DETAILED DESCRIPTION:
Eligible patients will be randomly assigned to either the investigational treatment arm (RB alternating with RBAC) or the standard treatment arm (RB) in a 1:1 ratio. Patients will be stratified by age (≥70 years vs. 60-69), histologic morphology (blastoid/pleomorphic vs. non-blastoid/non-pleomorphic), and MIPI-C risk score (0/1 vs. 2/3).

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed, previously untreated, histologically confirmed CD20+ mantle cell lymphoma, confirmed by WHO classification criteria
2. age ≥70 years or 60-69 years if the patients are ineligible for high-dose therapy with autologous stem cell transplantation.
3. ECOG performance status 2 or less
4. Adequate organ functions

   * adequate heart function: LVEF ≥50% by echocardiography or MUGA
   * adequate renal function: serum creatinine ≤ 2.0mg/dL or CrCl ≥40 mL/min based on the Cockcroft-Gault method
   * adequate hepatic function: ≤2.5 times the upper limit of ALT (≤5 times the upper limit of ALT if the elevation is attributed by underlying lymphoma) and ≤2 times the upper limit of ALT (≤3 times the upper limit of total bilirubin if the elevation is attributed by underlying lymphoma)
   * adequate hematologic function: absolute neutrophil counts (ANC) ≥ 1,500/mL, platelet counts ≥ 100,000/mL (any ANC and platelet counts are allowed, if they were related to bone marrow involvement)
5. Written informed consent

Exclusion Criteria:

1. In-situ mantle cell lymphoma
2. Ann Arbor stage 1 disease
3. Prior treatment for Hodgkin lymphoma or non-Hodgkin lymphoma within the last 5 years.
4. Active malignancy within the past 3 years except for localized non-melanoma skin cancer, papillary thyroid cancer, cervical carcinoma in situ, breast cancer in situ, or localized prostate cancer that has been definitely treated,
5. Central nervous system involvement
6. HBsAg (+) or anti-HBc Ab (+) (patients will be eligible if they receive appropriate prophylactic antiviral therapy using entecavir, tenofovir, and so on)
7. History of prior hepatitis C infection (patients positive for HCV IgG will be eligible if they are negative for HCV-RNA)
8. Known history of human immunodeficiency virus (HIV) infection
9. any serious illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study

   * Congestive heart failure ≥ NYHA class 3
   * Acute coronary syndrome within 6 months (unstable angina or new-onset angina, myocardial infarct, or ventricular arrhythmia)
   * History of significant neurological or psychological disorder including dementia and seizure disorder
   * Severe chronic obstructive pulmonary disease with hypoxemia
   * Cerebrovascular disease including transient ischemic attack within the past 6 months
   * Non-healing wound, ulcer, or bone fracture
   * Active uncontrolled bacterial, viral, or fungal infection requiring systemic therapy
10. concomitant administration of any other experimental drugs under investigation
11. Known hypersensitivity to bendamustine, rituximab, cytarabine, or mannitol
12. major surgical procedure or significant trauma within 28 days before start of study treatment, open biopsy within 7 days before start of study treatment
13. If the patient's partner is a woman who could possibly get pregnant, men who didn't have a vasectomy must agree to use medically recommended methods for adequate contraception (tubal ligation, intrauterine devices, or barriers [diaphragm, cervical cap] in the patient's partner and the use of condoms in men) when sexually active.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-freesurvival | Up to 84 months

SECONDARY OUTCOMES:
Overall Survival | Up to 84 months
Duration of Response | Up to 84 months
Event Free Survival | Up to 84 months
Overall response rate | Up to 84 months
Adverse events | From the day 1 of the clinical trial to 28 days after last drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No